CLINICAL TRIAL: NCT03326076
Title: Evaluation of Patient Outcomes From the Kidney Allograft Outcomes AlloSure Registry
Acronym: KOAR
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: CareDx (Industry)
Responsible Party: Sponsor
Other Study IDs: KOAR
Record Dates: First submitted 2017-10-24; First posted 2017-10-30 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Kidney Transplant Rejection
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma from venous blood will be collected and cell-free DNA will be extracted from the plasma for analysis of donor-derived cell-free DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Primary donor-derived cell-free DNA: 300 patients with planned renal surveillance biopsies at 12 months post-transplantation
  Interventions: Diagnostic Test: Donor-derived cell-free DNA (AlloSure®)
- Control: A matched control cohort of 1000 patients with planned renal surveillance biopsies at 12 months post-transplantation but were not managed with donor-derived cell-free DNA (AlloSure®) or KidneyCare will be retrospectively selected
  Interventions: Other: Standard care
- Secondary donor-derived cell-free DNA: 1200 patients without planned renal surveillance biopsies at 12 months post-transplantation
  Interventions: Diagnostic Test: Donor-derived cell-free DNA (AlloSure®)
- Primary KidneyCare®: 300 patients with planned renal surveillance biopsies at 12 months post-transplantation
  Interventions: Diagnostic Test: Donor-derived cell-free DNA (AlloSure®); Diagnostic Test: Peripheral blood gene expression profiling (AlloMap Kidney); Diagnostic Test: Analytic platform (IBox)
- Secondary KidneyCare®: 1200 patients without planned renal surveillance biopsies at 12 months post-transplantation
  Interventions: Diagnostic Test: Donor-derived cell-free DNA (AlloSure®); Diagnostic Test: Peripheral blood gene expression profiling (AlloMap Kidney); Diagnostic Test: Analytic platform (IBox)

INTERVENTIONS:
Diagnostic Test: Donor-derived cell-free DNA (AlloSure®) — Patients will receive donor-derived cell-free DNA testing for surveillance and for-cause. The planned surveillance will occur at months 1, 2, 3, 4, 6, 9, and 12 post-transplant and quarterly in year 2 and year 3.
  Groups: Primary KidneyCare®; Primary donor-derived cell-free DNA; Secondary KidneyCare®; Secondary donor-derived cell-free DNA
Other: Standard care — Current standard methods for monitoring of renal allograft recipients for rejection (e.g. donor-specific antibodies, serum creatinine, proteinuria, renal allograft biopsy)
  Groups: Control
Diagnostic Test: Peripheral blood gene expression profiling (AlloMap Kidney) — Patients will receive peripheral blood gene expression profiling testing for surveillance and for-cause. The planned surveillance will occur at months 1, 2, 3, 4, 6, 9, and 12 post-transplant and quarterly in year 2 and year 3.
  Groups: Primary KidneyCare®; Secondary KidneyCare®
Diagnostic Test: Analytic platform (IBox) — Patients will receive IBox testing for surveillance and for-cause. The planned surveillance will occur at months 1, 2, 3, 4, 6, 9, and 12 post-transplant and quarterly in year 2 and year 3.
  Groups: Primary KidneyCare®; Secondary KidneyCare®

SUMMARY:
This is an observational study to evaluate safety and efficacy outcomes in renal transplant recipients in whom post-transplant care is managed using AlloSure®. AlloSure® is a non-invasive test to measure donor-derived cell-free DNA (dd-cfDNA). The AlloSure test is intended to assess the probability of allograft rejection in kidney transplant recipients with clinical suspicion of rejection and to inform clinical decision-making regarding the necessity of renal biopsy in such patients at least 2 weeks post-transplant in conjunction with standard clinical assessment.

Amendment 1 (A1): Is an observational study to develop and validate the clinical use of KidneyCare®.

DETAILED DESCRIPTION:
The AlloSure test has been approved for Medicare coverage for clinical use when a physician determines there is a need to assess the probability of allograft rejection in kidney transplant recipients. The DART study suggests that use of the non-invasive AlloSure test to measure donor-derived cell-free DNA (dd-cfDNA) can be used to discriminate active rejection in a renal transplant recipient. Use of the test may reduce invasive percutaneous renal biopsy procedures among patients with a suspicion of rejection.

Amendment 1 (A1) is intended to enable the development of KidneyCare® which is a panel test which includes the clinically validated commercial AlloSure dd-cfDNA test, combined with AlloMap Kidney which is a peripheral blood gene expression profiling test currently under development, and iBox, which is an analytic platform that predicts allograft survival at 3, 5, 7 and 10 years using a proprietary software algorithm based on a number of clinical inputs. The AlloMap Kidney and the iBox components are not yet clinically validated and so will not be used for patient management and are being developed through this study.

ELIGIBILITY:
KOAR Inclusion Criteria:

1. Patient's health care provider adopts and intends to apply the center's AlloSure Routine Testing Schedule as part of the information used to manage the patient.
2. Subjects willing to provide written informed consent to participate.

KOAR Exclusion Criteria:

___________________________________________________________

Exclusions for AlloSure® Intended Use

Specimens from patients for whom any of the following are true will not be tested:

1. Recipients of transplanted organs other than kidney
2. Recipients of a transplant from a monozygotic (identical)
3. Recipients of a bone marrow transplant
4. Recipients who are pregnant
5. Recipients who are under the age of 18
6. Recipient who are less than 14 days post-transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All eligible renal transplant recipients who meet the inclusion/exclusion criteria will be a part of this observational study.
  The control cohort will include the patients cared for without the use of AlloSure® or KidneyCare at the participating centers who received their transplant in the 6 months prior to the enrollment start for the primary cohort.
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2018-01-23 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Interstitial fibrosis/tubular atrophy (IF/TA) quantified by Banff Working Group biopsy grade(s) at 12 months post-transplant in AlloSure® and renal allograft biopsy managed patients | Feb-2020
Total number of biopsies planned and performed post-transplant, including both surveillance and clinically indicated biopsies | Feb-2020

SECONDARY OUTCOMES:
Transplant glomerulopathy (TG) | Dec-2022
  Evaluated at one-year post-transplant, quantified by biopsy-based histopathology grade(s)
Patient and graft survival | Dec-2022
  Evaluated at years 1, 2, and 3 post-transplant
Serum creatinine | Dec-2022
  Evaluated at years 1, 2, and 3 post-transplant
Estimated glomerular filtration rate | Dec-2022
  Evaluated at years 1, 2, and 3 post-transplant
Sensitivity of AlloSure for active rejection | Dec-2022
Specificity of AlloSure for active rejection | Dec-2022
Negative Predictive Value (NPV) of AlloSure for active rejection | Dec-2022
Positive Predictive Value (PPV) of AlloSure for active rejection | Dec-2022
Develop and validate the clinical use of KidneyCare® | Dec-2022

CONTACTS AND LOCATIONS:
Locations (72):
- United States (72):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Loma Linda Medical Center, Loma Linda, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of Southern California, Los Angeles, California
  - University of California, Los Angeles, Los Angeles, California
  - Stanford Health Care, Palo Alto, California
  - UC Davis Medical Center, Sacramento, California
  - California Pacific Medical Center, San Francisco, California
  - University of California San Francisco, San Francisco, California
  - University of Colorado Hospital, Aurora, Colorado
  - University of Colorado- Anschutz Medical Campus, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - Georgetown University, Washington D.C., District of Columbia
  - George Washington University, Washington D.C., District of Columbia
  - University of Miami/Jackson Memorial Hospital, Miami, Florida
  - AdventHealth, Orlando, Florida
  - Tampa General Hospital, Tampa, Florida
  - Cleveland Clinic - Weston, Weston, Florida
  - Augusta University, Augusta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Loyola University, Maywood, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky Chandler Hospital, Lexington, Kentucky
  - Tulane University Medical Center, New Orleans, Louisiana
  - Ochsner Foundation Hospital, New Orleans, Louisiana
  - Willis-Knighton Physician Network/ John C. McDonald Regional Transplant Center, Shreveport, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - The University of Missouri, Columbia, Missouri
  - Washington University (Barnes Jewish Hospital), St Louis, Missouri
  - Washington University, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Saint Barnabus Medical Center, Livingston, New Jersey
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Erie County Medical Center, Buffalo, New York
  - Montefiore Medical Center, The Bronx, New York
  - Metrolina Nephrology Associates, Charlotte, North Carolina
  - Duke University, Durham, North Carolina
  - East Carolina University/Vidant Medical Center, Greenville, North Carolina
  - Wake Forest Baptist Medical Center- Department of General Surgery, Winston-Salem, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - The Oklahoma Transplant Center at OU Medical Center, Oklahoma City, Oklahoma
  - Integris Baptist Medical Center, Oklahoma City, Oklahoma
  - Geisinger Clinic, Danville, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Methodist Healthcare Foundation, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - UT Southwestern, Dallas, Texas
  - Baylor All Saints Medical Center, Fort Worth, Texas
  - Texas Research Institute, Fort Worth, Texas
  - Houston Methodist Hospital, Houston, Texas
  - UT Health San Antonio, San Antonio, Texas
  - Baylor Scott & White Medical Center, Temple, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Utah, Salt Lake City, Utah
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - Sacred Heart Medical Center, Spokane, Washington

REFERENCES:
- [Background] Bloom RD, Bromberg JS, Poggio ED, Bunnapradist S, Langone AJ, Sood P, Matas AJ, Mehta S, Mannon RB, Sharfuddin A, Fischbach B, Narayanan M, Jordan SC, Cohen D, Weir MR, Hiller D, Prasad P, Woodward RN, Grskovic M, Sninsky JJ, Yee JP, Brennan DC; Circulating Donor-Derived Cell-Free DNA in Blood for Diagnosing Active Rejection in Kidney Transplant Recipients (DART) Study Investigators. Cell-Free DNA and Active Rejection in Kidney Allografts. J Am Soc Nephrol. 2017 Jul;28(7):2221-2232. doi: 10.1681/ASN.2016091034. Epub 2017 Mar 9. PMID 28280140
- [Background] Grskovic M, Hiller DJ, Eubank LA, Sninsky JJ, Christopherson C, Collins JP, Thompson K, Song M, Wang YS, Ross D, Nelles MJ, Yee JP, Wilber JC, Crespo-Leiro MG, Scott SL, Woodward RN. Validation of a Clinical-Grade Assay to Measure Donor-Derived Cell-Free DNA in Solid Organ Transplant Recipients. J Mol Diagn. 2016 Nov;18(6):890-902. doi: 10.1016/j.jmoldx.2016.07.003. Epub 2016 Oct 7. PMID 27727019